CLINICAL TRIAL: NCT00995579
Title: Assessment of Energy Expenditure by Indirect Calorimetry for a Daily 10,000 Steps Goal
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Liying Wang, School and Graduate Institute of Physical Therapy, National Taiwan University
Other Study IDs: 200809081R
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Physical Activity; Energy Expenditure
Keywords: Physical Activity; Energy Expenditure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy college volunteers

SUMMARY:
The purpose of this study was to measure the actual energy expenditure (EE) using indirect calorimetry for the 10,000 steps goal, and compared to the estimated EE using predictive equation.

DETAILED DESCRIPTION:
Physical inactivity is considered a major risk factor for a number of adverse health outcomes such as obesity, hypertension, cardiovascular disease, diabetes mellitus, and all-cause mortality. Certain guidelines specifically recommend taking 10,000 steps per day for a goal. Some of pedometers have a function of energy expenditure estimation in addition to counting steps. However, the EE derived from pedometers is the indirect estimation calculated from metabolic calculations instead of direct measurement.The purpose of this study was to measure the actual energy expenditure (EE) using indirect calorimetry for the 10,000 steps goal, and compared to the estimated EE using predictive equation.

Twenty healthy college volunteers were recruited. First, height and weight were measured from each subject. Body mass index (BMI) was calculated as the ratio of weight to height in meters squared. We used BioScan 920 to get all subjects' body composition data including fat mass and fat-free mass. Followed by measurements of basic characteristics, all subjects wore the pedometer and walked 10,000 steps on the treadmill. The walking speeds ranged from 3.0 to 4.0 miles per hour (mph) according to different gender. The speed of 4.0 mph was set for male and 3.0 mph was set for female. If the subject could'nt follow the pre-set speed, he/she could walk with self-comfortable speed but the speed should be in the range of 3.0 to 4.0 mph defined as moderate intensity of ACSM's recommendation. Subjects rested on the chair with back support for 3 minutes and then completed the 10,000 steps goal. After recovery for 3 minutes, the data collection was finished. The stopping criteria of the test were as follows: dizziness, nausea, dyspnea, or leg fatigue which leads subjects unable to continue. Expired gas was collected using the Cosmed K4b2 portable indirect calorimetry system, and EE was monitored breath-by-breath according to the following formula:

EE (Kcal/min)= 3.781×VO2＋1.237×VCO2

where VO2 represents the standardized oxygen consumption per minute, and VCO2 is the carbon dioxide production per minute. Estimated EE was calculated by the predictive equation published by ACSM:

VO2 (ml/kg/min)= 0.1×S (m/min)＋1.8×S×G (%)＋3.5

where S represents the walking speed, and G is the walking grade.

The total walking duration and distance for taking 10,000 steps were also recorded. Pulmonary function tests were performed on the other day to get each subject's functional vital capacity (FVC). We used this parameter to estimate subject's predicted maximal minute ventilation (predicted max VE) according to the equation provided in the guidelines of American Thoracic Society (ATS) for cardiopulmonary exercise testing:

VE (L/min)= 26.3×VC-34

where VC represents vital capacity. The ratio of averaged VE during walking and predicted maximal VE was calculated to determine the level of exercise intensity for taking 10,000 steps.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 y/o

Exclusion Criteria:

* Unstable systemic disease, respiratory diseases, cardiac diseases or other clinical diagnosis which would affect outcome measure
* Subjects who answered yes to any of the PAR-Q questions or who were not physically able to complete the test

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy college volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
energy expenditure | 3 months

SECONDARY OUTCOMES:
Body composition: fat mass and fat-free mass | 3 months
Pulmonary function: FVC, FEV1, FEV1/FVC | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Liying Wang, Ph.D., Principal Investigator — chool and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan